CLINICAL TRIAL: NCT00095082
Title: Efficacy and Safety Comparison of Insulin Detemir Plus Insulin Aspart Versus Insulin Glargine Plus Insulin Aspart in Type 1 Diabetes
Brief Title: Safety and Efficacy of Insulin Detemir Plus Insulin Aspart Against Insulin Glargine Plus Insulin Aspart as Mealtime Insulin in Type 1 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN304-1430; 2004-000086-35 (EudraCT Number)
Record Dates: First submitted 2004-10-29; First posted 2004-11-01 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
Keywords: Diabetes Mellitus, Type I
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin Detemir; Insulin Glargine; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: insulin detemir
Drug: insulin glargine
Drug: insulin aspart

SUMMARY:
This trial is conducted in Europe and the United States of America (USA). The purpose of this study is to test whether insulin detemir is a safe and at least as effective alternative to insulin glargine for the control of blood glucose in basal/bolus therapy in patients with type I diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes for at least 12 months
* Current treatment with basal-bolus insulin regimen for more than or equal to 3 months
* HbA1c less than or equal to 11.0%

Exclusion Criteria:

* Proliferative retinopathy or maculopathy
* Recurrent major hypoglycaemia
* Impaired hepatic or renal function
* Cardiac problems or uncontrolled hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 447 (Actual)
Dates: Start 2004-09; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
HbA1c | after 1 year trial period

SECONDARY OUTCOMES:
Adverse events
Body weight
Hypoglycemia
Blood glucose
Insulin Treatment Satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (77):
- United States (27):
  - Novo Nordisk Investigational Site, Anaheim, California
  - Novo Nordisk Investigational Site, Huntington Beach, California
  - Novo Nordisk Investigational Site, Inglewood, California
  - Novo Nordisk Investigational Site, Irvine, California
  - Novo Nordisk Investigational Site, La Jolla, California
  - Novo Nordisk Investigational Site, Hollywood, Florida
  - Novo Nordisk Investigational Site, Jacksonville, Florida
  - Novo Nordisk Investigational Site, Lake Mary, Florida
  - Novo Nordisk Investigational Site, Melbourne, Florida
  - Novo Nordisk Investigational Site, Tampa, Florida
  - Novo Nordisk Investigational Site, Vero Beach, Florida
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Idaho Falls, Idaho
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Topeka, Kansas
  - Novo Nordisk Investigational Site, Hyattsville, Maryland
  - Novo Nordisk Investigational Site, Detroit, Michigan
  - Novo Nordisk Investigational Site, St Louis, Missouri
  - Novo Nordisk Investigational Site, Omaha, Nebraska
  - Novo Nordisk Investigational Site, Las Vegas, Nevada
  - Novo Nordisk Investigational Site, Berlin, New Jersey
  - Novo Nordisk Investigational Site, Sea Girt, New Jersey
  - Novo Nordisk Investigational Site, Asheville, North Carolina
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
- Finland (5):
  - Novo Nordisk Investigational Site, Helsinki
  - Novo Nordisk Investigational Site, Kuopio
  - Novo Nordisk Investigational Site, Oulu
  - Novo Nordisk Investigational Site, Pori
  - Novo Nordisk Investigational Site, Vantaa
- France (7):
  - Novo Nordisk Investigational Site, Angers
  - Novo Nordisk Investigational Site, Antibes
  - Novo Nordisk Investigational Site, Brest
  - Novo Nordisk Investigational Site, Grenoble
  - Novo Nordisk Investigational Site, La Rochelle
  - Novo Nordisk Investigational Site, Mougins
  - Novo Nordisk Investigational Site, Toulouse
- Germany (15):
  - Novo Nordisk Investigational Site, Alsdorf
  - Novo Nordisk Investigational Site, Bad Kreuznach
  - Novo Nordisk Investigational Site, Dormagen
  - Novo Nordisk Investigational Site, Dresden
  - Novo Nordisk Investigational Site, Flensburg
  - Novo Nordisk Investigational Site, Friedrichsthal
  - Novo Nordisk Investigational Site, Genthin
  - Novo Nordisk Investigational Site, Hamburg
  - Novo Nordisk Investigational Site, Herrenberg
  - Novo Nordisk Investigational Site, Kippenheim
  - Novo Nordisk Investigational Site, Rehlingen-Siersburg
  - Novo Nordisk Investigational Site, Saint Ingbert
  - Novo Nordisk Investigational Site, Speyer
  - Novo Nordisk Investigational Site, Völklingen
  - Novo Nordisk Investigational Site, Würzburg
- Netherlands (6):
  - Novo Nordisk Investigational Site, Almere Stad
  - Novo Nordisk Investigational Site, Apeldoorn
  - Novo Nordisk Investigational Site, Capelle aan den IJssel
  - Novo Nordisk Investigational Site, Dordrecht
  - Novo Nordisk Investigational Site, Leeuwarden
  - Novo Nordisk Investigational Site, Zoetermeer
- Sweden (5):
  - Novo Nordisk Investigational Site, Norrköping
  - Novo Nordisk Investigational Site, Örebro
  - Novo Nordisk Investigational Site, Stockholm
  - Novo Nordisk Investigational Site, Umeå
  - Novo Nordisk Investigational Site, Vaxjo
- United Kingdom (12):
  - Novo Nordisk Investigational Site, Abergavenny
  - Novo Nordisk Investigational Site, Ayr
  - Novo Nordisk Investigational Site, Brighton
  - Novo Nordisk Investigational Site, Bristol
  - Novo Nordisk Investigational Site, Cosham
  - Novo Nordisk Investigational Site, Dundee
  - Novo Nordisk Investigational Site, Glasgow
  - Novo Nordisk Investigational Site, Livingstone
  - Novo Nordisk Investigational Site, Plymouth
  - Novo Nordisk Investigational Site, Sheffield
  - Novo Nordisk Investigational Site, Watford
  - Novo Nordisk Investigational Site, Wirral, Merseyside

REFERENCES:
- [Result] Heller S, Koenen C, Bode B. Comparison of insulin detemir and insulin glargine in a basal-bolus regimen, with insulin aspart as the mealtime insulin, in patients with type 1 diabetes: a 52-week, multinational, randomized, open-label, parallel-group, treat-to-target noninferiority trial. Clin Ther. 2009 Oct;31(10):2086-97. doi: 10.1016/j.clinthera.2009.10.006. PMID 19922879
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com